CLINICAL TRIAL: NCT04462302
Title: Internet-delivered Management of Pain Among Cancer Treatment Survivors
Brief Title: An Internet-based Program to Help Cancer Survivors Manage Pain
Acronym: IMPACTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00066906; 3UG1CA189824-06S1 (NIH); WF-1901 (Other: Wake Forest NCORP Research Base); NCI-2020-02315 (Registry Identifier: NCI CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Cancer pain; Survivor; Pain; Pain coping
MeSH Terms: conditions — Neoplasms; Cancer Pain; Pain

STUDY DESIGN:
Intervention Model Description: This is a parallel group randomized controlled, prospective study that examines the effect of an Internet-based pain coping skills program on pain severity and pain interference among adult cancer survivors experiencing persistent cancer-related pain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based program + Pain Education (Experimental): If you are in this group, in additional to your usual care, you will be provided access to the 8-session Internet-based pain program plus pain education. You will need to complete your sessions within 10 weeks of being provided your log-in code. You will be allowed to revisit sessions that you have completed during this 10 weeks. After completion of the study, you will still be provided access to the 8-session Internet-based pain program.
  Interventions: Behavioral: Internet-based pain coping skills program
- Pain Education Only (No Intervention): If you are in this group, in addition to your usual care, you will be provided pain education at your initial clinic visit. After you have completed the 6-month follow up assessment, you will be provided a secure log-in code and invited to complete the 8 sessions of this Internet-based pain program on your own.

INTERVENTIONS:
Behavioral: Internet-based pain coping skills program — The purpose of this study is to determine if an 8-session Internet-based pain management program can help you better manage your cancer-related pain.
  Arms: Internet-based program + Pain Education

SUMMARY:
To determine whether an Internet-based pain coping skills program plus enhanced usual care, compared to enhanced usual care alone, yields significant improvements in the co-primary outcomes of pain severity (as measured by the Brief Pain Inventory (BPI)) and pain interference (also measured by the BPI) from baseline to the post-intervention assessment for cancer survivors with persistent pain.

DETAILED DESCRIPTION:
This is a parallel group randomized controlled, prospective study that examines the effect of an Internet-based pain coping skills program on pain severity and pain interference among adult cancer survivors experiencing persistent cancer-related pain. The study also explores the effects of an Internet-based pain coping skills program on opioid/analgesic medication use, health-related quality of life, pain management self-efficacy and various other factors relevant among populations with persistent pain (i.e., fatigue, sleep, emotional distress, positive affect, pain impact, perceived cognitive problems, and cognitive performance), as well as qualitative assessments of participants experiences with pain and the intervention. A total of 250 participants will be enrolled (125 per arm) and randomized into the internet program arm (plus enhanced usual care) or Enhanced Usual Care alone.

Each participant will be enrolled in the study for 9 months (from randomization at week 0 to the final follow-up assessment at week 34).

ELIGIBILITY:
Inclusion Criteria:

Must have a documented diagnosis of invasive cancer that has been treated with either single modality therapy or any combination of surgery, radiation, and chemotherapy/drug therapy (e.g. cytotoxic therapy, targeted therapy, immunotherapy, hormonal therapy, etc.). Patients with a cancer history of only superficial skin cancers or in situ malignancy are not eligible.

* May be either off all treatment OR actively receiving anticancer therapy in an adjuvant setting, maintenance setting, or for active cancer.

  * Patients who currently undergoing anticancer therapy should not have any plans to change or adjust their treatment during the intervention period. This includes changing to another therapy or ending therapy entirely.
  * Patients who are currently receiving anticancer therapy at the screening process must have been on current therapy for at least four weeks. Alternatively, if they are planning to discontinue therapy before enrolling, they must have been off therapy for four weeks prior to enrollment.
  * A minimum of four weeks must have elapsed since the most recent MAJOR surgical intervention.
  * A minimum of two weeks must have elapsed since the most recent MINOR surgical procedure (e.g., port placement).
  * In addition, eligible patients must not have a planned surgical procedure or course of radiation therapy during the 3-month study intervention period (i.e., the three months leading up to primary outcome evaluation-timepoint.
* Patients who are no longer receiving anticancer therapy must be less than/equal to 5 years since the completion of their anticancer therapy (e.g., time since the last day of chemotherapy administration, time since last day of radiotherapy, etc.).
* Must have pain indicated by a score of ≥ 4 on PROMIS Pain Intensity (1a) scale, using the Pain Eligibility Interview.
* Must have a score of "Most Days" or higher on the Graded Chronic Pain Scale Revised (Abbreviated) using the Pain Eligibility Interview.
* Patients do not have to be on analgesic medications of any kind in order to participate. If they are taking analgesics, they must be on a stable analgesic regimen (i.e., no changes to the prescribed analgesic regimen) over a period of at least 14 days prior to enrollment. Eligible patients should not have planned upward dose titration of their analgesics during the 3-month study intervention period (i.e., the three months leading up to primary outcome evaluation timepoint. Patients may elect to decrease their analgesic use during the study as per discussions with their provider. Unexpected dose adjustments including dose escalations as a result of unforeseen clinical need is allowed in all patients at all times during the study. Cannabis prescribed for medicinal purposes would qualify as an analgesic in this context.
* Must have pain of new onset or significantly exacerbated since the time of cancer diagnosis or initiation of cancer treatment
* Must be expected to be able to complete all study activities including the 22- and 34-week follow-up assessments according to the treating/referring clinician (e.g., treating clinician feels the patient is unlikely to develop progressive disease requiring additional active cancer therapy through the 6-month follow-up period).
* ECOG performance status of 0, 1, or 2.
* Age ≥18 years at the time of study entry
* Must be able to speak, read and understand English.

Exclusion Criteria:

* Has a disability that precludes completion of study activities (e.g., severe vision or hearing impairment, diagnosis of dementia or clinical evidence of severe cognitive impairment, diagnosis or clinical evidence of severe psychiatric disorder, or diagnosed drug or alcohol abuse disorder), as per patient report or documented in the medical record.
* Reports only preexisting pain conditions unrelated to cancer or cancer treatment (e.g., migraine or tension headache, arthritis, back disorders, bursitis/tendonitis, injuries, fibromyalgia).
* Has a known or suspected diagnosable substance use disorder or opioid overuse disorder (according to DSM-5 criteria), or is actively receiving treatment for a substance use disorder, as per patient report or documented in the medical record.
* Currently being prescribed buprenorphine or suboxone.
* Patients enrolled on hospice care or end-of-life palliative care are not eligible for enrollment. Patients whose local care network provides an opportunity for palliative (symptom management) or supportive care concurrent with active treatment following diagnosis (i.e. not solely as a palliative or end-of-life measure) are considered eligible for this study.
* Does not have reliable access to Internet or sufficient personal data plan, and is not willing to participate in the Tablet Lending Program provided for this study.
* Does not have a working email address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | Change from Baseline to 10 week
  The Pain Severity via Brief Pain Inventory (BPI) subscale score is the mean of 4 items measuring current pain, pain on average, and pain at its worst and least in the past 7 days on a scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain Interference | Change from Baseline to 10 week
  The Pain Interference via Brief Pain Inventory (BPI) subscale score is the mean rating of 7 items measuring impact of pain on walking, work, mood, enjoyment of life, relations with others, sleep, general activity on a scale from 0 (does not interfere) to 10 (completely interferes).

SECONDARY OUTCOMES:
Pain Severity | 22 and 34 weeks
  The Pain Severity via Brief Pain Inventory (BPI) subscale score is the mean of 4 items measuring current pain, pain on average, and pain at its worst and least in the past 7 days on a scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain Interference | 22 and 34 weeks
  The Pain Interference via Brief Pain Inventory (BPI) subscale score is the mean rating of 7 items measuring impact of pain on walking, work, mood, enjoyment of life, relations with others, sleep, general activity on a scale from 0 (does not interfere) to 10 (completely interferes).
Opioid/analgesic medication use | Baseline and 10 week
  A participant recall during clinic visits of typical daily medication use. This will be converted to morphine milligram equivalents (MME).
Opioid/analgesic medication use | Baseline, 10, 22, and 24 week
  7-day medication diaries to capture participants' use of all medications each day during a 7-day period. Self-reports will be converted to morphine milligram equivalents (MME).
Health-Related Quality of Life | Baseline, 10, 22, and 24 week
  Health-Related Quality of Life will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (Short Form-6b). The six items are summed to give a score from 6 to 30, with higher scores representing better physical function.
Pain Management Self-Efficacy | Baseline, 10, 22, and 24 week
  Pain Management Self-Efficacy will be assessed with the Chronic Pain Self-Efficacy Scale. The self-efficacy for pain management subscale (PSE) consists of five items summed to give a score from 50-500, the self-efficacy for physical function subscale (FSE) consists of nine items summed to give a score from 90-900, and the self-efficacy for coping with symptoms subscale (CSE) consists of eight items summed to give a score from 80-800. For all subscales, higher scores represent greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, MD, Study Chair — Wake Forest University Health Sciences
Locations (150):
- United States (149):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - John B. Amos Cancer Center, Columbus, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Carle BroMenn Outpatient Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Marshfield Medical Center Dickinson, Iron Mountain, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CentraState Medical Center, Freehold, New Jersey
  - Hackettstown Medical Center, Hackettstown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - Chilton Medical Center, Pompton, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest University at Lexington, Lexington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Peninsula Cancer Institute - Gloucester, Gloucester, Virginia
  - Peninsula Cancer Institute - Newport News, Newport News, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Peninsula Cancer Institute - Cancer Specialists of Tidewater, Virginia Beach, Virginia
  - Peninsula Cancer Institute - Williamsburg, Williamsburg, Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- FHP Health Center-Guam, Tamuning, GU, Guam

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu